CLINICAL TRIAL: NCT05899179
Title: A Multicenter, Randomized, Double-blind, Controlled Phase Ⅲ Trial of Recombinant Mycobacterium Tuberculosis Fusion Protein (EC) for the Diagnosis of Mycobacterium Tuberculosis Infection in 65-year-olds and Above
Brief Title: Clinical Study of Recombinant Mycobacterium Tuberculosis Fusion Protein for 65-year-olds and Above
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: LKM-2022-EC01
Record Dates: First submitted 2023-04-11; First posted 2023-06-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: Latent Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis | interventions — Tuberculin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left arm injection EC group (Experimental): The Recombinant Mycobacterium tuberculosis fusion protein(EC) was injected intradermally into the volar side of the left forearm by the Mondu's method. After observing no abnormality for 5 minutes, TB-PPD was injected intradermally into the volar side of the right forearm.
  Interventions: Biological: Recombinant Mycobacterium Tuberculosis Fusion Protein; Biological: Purified Protein Derivative of Tuberculin
- Right arm injection EC group (Active Comparator): The Recombinant Mycobacterium tuberculosis fusion protein(EC) was injected intradermally into the volar side of the right forearm by the Mondu's method. After observing no abnormality for 5 minutes, TB-PPD was injected intradermally into the volar side of the left forearm.
  Interventions: Biological: Recombinant Mycobacterium Tuberculosis Fusion Protein; Biological: Purified Protein Derivative of Tuberculin

INTERVENTIONS:
Biological: Recombinant Mycobacterium Tuberculosis Fusion Protein — Dosage form:injection. Main ingredients and contents: Recombinant Mycobacterium tuberculosis fusion protein, 0.3ml, 0.5ml, 1.0ml per bottle.
  1. This product is used alone: 0.1ml (5U) of this product is inhaled and injected into the palmar skin of the forearm by the Mondu's method. 2. This product combined with TB-PPD: 0.1ml(5U) of this product and 0.1ml(5U) of TB-PPD were inhaled respectively, and the product was injected intradermally into the volar side of the left forearm by the Mondu's method. After observing no abnormality for 5 minutes, TB-PPD was injected intradermally into the volar side of the right forearm.
  Other Names: EC
Biological: Purified Protein Derivative of Tuberculin — Dosage form:injection. Main ingredients and contents:Pure protein derivatives of tuberculin,0.1ml per bottle.
  Usage:0.1ml (5IU) of this product is inhaled and injected into the palmar skin of the forearm by the Mondu's method.
  Other Names: TB-PPD

SUMMARY:
A multicenter, randomized, blind, controlled trial design was used to select 240 tuberculosis (TB) patients, 120 non-tuberculous community population with other lung diseases, and 420 healthy community population without other lung diseases who met the inclusion criteria of this study. Blood supply specific gamma-interferon (T-SPOT) detection was performed first. Then, EC and Purified Protein derivation of tuberculin (TB-PPD) skin tests were performed on both arms, and the recorded results were observed. The first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases were included in the trial subgroup. Physical examination, blood routine, urine routine, liver and kidney function, and electrocardiogram tests were required before and 7 days after skin test after study number assignment.

DETAILED DESCRIPTION:
A multicenter, randomized, blind, controlled trial design was adopted in this study. Subjects were enrolled in this clinical study after being qualified by physical examination, vital signs detection (body temperature, blood pressure, pulse and respiration), chest imaging (DR/CT) examination, mycobacterium tuberculosis etiology examination, HIV antibody detection, fasting blood glucose detection, etc.

A total of 240 TB patients, 120 non-tuberculous community people with other lung diseases, and 420 healthy community people without other lung diseases were selected for inclusion in this study. Blood samples were collected for specific gamma-interferon (T-SPOT) detection, and then EC and TB-PPD in the same double arm skin test were used to observe and record the results.

The first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases were included in the trial subgroup. Physical examination, blood routine, urine routine, liver and kidney function, and electrocardiogram tests were required before and 7 days after skin test after study number assignment.

Vital signs (body temperature, blood pressure, pulse and respiration) were measured 30min and 24h after skin test, and body temperature was measured 48h and 72h after skin test. The skin reaction at the injection site was observed at 0min, 24h, 48h and 72h after skin test.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old and above (≥ 65 years old), male or female, the subjects themselves voluntarily participate in this study, sign the informed consent form, and can understand and comply with the requirements of the trial protocol to participate in follow-up.
* Normal underarm body temperature (< 37.3 °C);
* Tuberculosis patients: pulmonary tuberculosis patients and extrapulmonary tuberculosis patients diagnosed by researchers as confirmed cases of tuberculosis and clinically diagnosed cases. Refer to the "WS288-2017 Tuberculosis Diagnostic Criteria" to formulate the diagnostic criteria for pulmonary tuberculosis in this protocol, see Annex 1 for details; The diagnostic criteria for extrapulmonary tuberculosis were formulated with reference to the Technical Guidelines for Tuberculosis Prevention and Control in China (2021 edition of the Chinese Center for Disease Control and Prevention), as detailed in Annex 2.
* Non-tuberculous community population with other lung diseases: there is a clear lung disease, but the study physician can exclude pulmonary tuberculosis based on the patient's clinical manifestations, chest imaging and laboratory tests. Diagnostic criteria for their main types of nontuberculous other lung diseases can be found in Annex 3;
* Community healthy people without other lung diseases: those who have no history of tuberculosis, no suspicious symptoms of tuberculosis, no history of respiratory tract and recent respiratory symptoms, and no obvious abnormalities in both lungs on chest imaging (DR) examination; After consultation, there is no history of heart, liver, kidney, digestive tract, nervous system, or psychiatric abnormalities.

Exclusion Criteria:

* Combined with the following serious diseases, such as advanced tumors, acute exacerbation of chronic obstructive pulmonary disease, acute or progressive liver disease or kidney disease, decompensated stage of congestive heart failure, autoimmune diseases (except those who do not need to use immune agents in the stable period), primary immunodeficiency diseases, etc.;
* Those suffering from acute infectious diseases (such as measles, pertussis, influenza, pneumonia, etc.), acute conjunctivitis, acute otitis media, extensive skin diseases and allergies;
* Those with known or suspected (or high-risk occurrence possibility) immune impairment or abnormalities, such as those receiving immunosuppressants or immune booster therapy, receiving glucocorticoids, immunoglobulin preparations other than the gastrointestinal tract or blood products or plasma extracts within 1 month;
* Those who have positive human immunodeficiency virus (HIV) antibody test results;
* Those who are participating in other new drug clinical trials or have participated in any other new drug clinical trials within 3 months before this clinical trial;
* Fasting blood glucose ≥ 10mmol/L after drug control;
* Blood pressure range: systolic blood pressure ≥ 180 mmHg and (or) diastolic blood pressure ≥ 110 mmHg (those who take drugs are uncontrollable);
* Any situation that the investigator believes is poor adherence or may affect the evaluation of the trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Measure the diameter of redness or induration at the reaction site | The skin test was performed at 0 minute after injection.
  The diameter of redness or induration at the reaction site was measured with a scale at 0 minute after skin testing. Take the larger one of redness or induration as the measurement result. The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) below 5 mm at any point in time is negative. The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) of not less than 5 mm at any point in time is positive. Where there are blisters, necrosis, lymphangitis are strong positive reaction.
Measure the diameter of redness or induration at the reaction site | The skin test was performed at 24 hours after injection.
  The diameter of redness or induration at the reaction site was measured with a scale at 24 hours after skin testing. Take the larger one of redness or induration as the measurement result. The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) below 5 mm at any point in time is negative.The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) of not less than 5 mm at any point in time is positive. Where there are blisters, necrosis, lymphangitis are strong positive reaction.
Measure the diameter of redness or induration at the reaction site | The skin test was performed at 48 hours after injection.
  The diameter of redness or induration at the reaction site was measured with a scale at 48 hours after skin testing.Take the larger one of redness or induration as the measurement result. The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) below 5 mm at any point in time is negative. The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) of not less than 5 mm at any point in time is positive. Where there are blisters, necrosis, lymphangitis are strong positive reaction.
Measure the diameter of redness or induration at the reaction site | The skin test was performed at 72 hours after injection.
  The diameter of redness or induration at the reaction site was measured with a scale at 72 hours after skin testing.Take the larger one of redness or induration as the measurement result. The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) below 5 mm at any point in time is negative. The average diameter of the reaction (sum of transverse and longitudinal diameters divided by 2) of not less than 5 mm at any point in time is positive. Where there are blisters, necrosis, lymphangitis are strong positive reaction.
Evaluate the incidence of all adverse events | Incidence of all adverse events within 7 days after injection.
  Incidence of all adverse events within 7 days after skin testing.
Evaluate the incidence of serious adverse event (SAE) | Incidence of SAE within 28 days after full vaccination
  Incidence of SAE within 28 days after injection
In subgroup, count the number of patients with changes in clinical significance of blood routine test before skin test compared with that 7 days after skin test | before injection
  The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases. In subgroup, venous blood was collected before skin test for blood routine (3ml) . The number of patients with changes in clinical significance of blood routine before skin test compared with that 7 days after skin test was counted.
In subgroup, count the number of patients with changes in clinical significance of urine routine test before skin test compared with that 7 days after skin test | before injection
  The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases.In subgroup, urine sample was collected before skin test for urine routine (10ml) .The number of patients with changes in clinical significance of urine routine test before skin test compared with that 7 days after skin test was counted.
In subgroup, count the number of patients with changes in clinical significance of liver and kidney function test before skin test compared with that 7 days after skin test | before injection
  The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases.In subgroup, venous blood was collected before skin test for liver and kidney function test (3ml) .The number of patients with changes in clinical significance of liver and kidney function test before skin test compared with that 7 days after skin test test was counted.
In subgroup, count the number of patients with changes in clinical significance of electrocardiogram test before skin test compared with that 7 days after skin test | before injection
  Electrocardiogram test was performed in subgroup before skin test . The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases .The number of patients with changes in clinical significance of electrocardiogram test before skin test compared with that 7 days after skin test was counted.
In subgroup, count the number of patients with changes in clinical significance of blood routine test 7 days after skin test compared with that before skin test | 7days after injection
  The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases. In subgroup, venous blood was collected 7 days after skin test for blood routine (3ml) . The number of patients with changes in clinical significance of blood routine test 7 days after skin test compared with that before skin test was counted.
In subgroup, count the number of patients with changes in clinical significance of urine routine test 7 days after skin test compared with that before skin test | 7days after injection
  The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases. In subgroup, urine sample was collected 7 days after skin test for urine routine (10ml) .The number of patients with changes in clinical significance of urine routine test 7 days after skin test compared with that before skin test was counted.
In subgroup, count the number of patients with changes in clinical significance of liver and kidney function test 7 days after skin test compared with that before skin test | 7days after injection
  The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases. In subgroup, venous blood was collected 7 days after skin test for liver and kidney function test (3ml) .The number of patients with changes in clinical significance of liver and kidney function test 7 days after skin test compared with that before skin test was counted.
In subgroup, count the number of patients with changes in clinical significance of electrocardiogram test 7 days after skin test compared with that before skin test | 7days after injection
  Electrocardiogram test was performed in subgroup. The subgroup included the first 24 cases of TB patients, the first 12 cases of non-tuberculous community population with other lung diseases, and the first 42 cases of healthy community population without other lung diseases 7 days after skin test.The number of patients with changes in clinical significance of electrocardiogram test 7 days after skin test compared with that before skin test was counted.

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, bachelor, Principal Investigator — Shenzhen Third People's Hospital
Locations (8):
- China (8):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Chest Hospital, Hefei, Anhui
  - Guangzhou Municipal Hospital of Chest Medicine, Guangzhou, Guangdong
  - The Third People's Hospital Of Shenzhen, Shenzhen, Guangdong
  - LiuZhou People's Hospital, Liuchow, Guangxi
  - Changsha Central Hospital, Changsha, Hunan
  - Wuxi NO.5 People's Hospital, Wuxi, Jiangsu
  - Wuhan Institute for Tuberculosis Control, Wuhan

IPD SHARING:
Plan to Share IPD: No